CLINICAL TRIAL: NCT02168335
Title: The Efficacy of OrasaltsTM in the Treatment of Gingivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Johannesburg (Other)
Responsible Party: Principal Investigator, Dr J. Pellow, Dr, University of Johannesburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DaSilva200814363; HDC01-35-2014 (Other: University of Johannesburg)
Record Dates: First submitted 2014-06-12; First posted 2014-06-20 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): OrasaltsTM
  1 level scoop of OrasaltsTM will be dissolved in warm water. Participants will rinse and gargle the mouth for 30 seconds, then expel and not swallow the mixture, twice daily
  Interventions: Other: OrasaltsTM
- Control group (Placebo Comparator): Sea salt
  1 level scoop of sea salt will be dissolved in warm water. Participants will rinse and gargle the mouth for 30 seconds, then expel and not swallow the mixture, twice daily
  Interventions: Other: Sea salt

INTERVENTIONS:
Other: OrasaltsTM — OrasaltsTM mouthwash is composed of 119.5g of natural sea salt, Arnica montana 30C, Echinacea angustifolia 30C, Staphysagria 30C, Phosphorus 30C, Hepar sulphuris 30C, 0.27g cinnamon and 0.27g of liquorice
  Arms: Treatment group
Other: Sea salt — Unmedicated sea salt
  Arms: Control group

SUMMARY:
Gingivitis is defined as inflammation of the gingiva. It is a common disease that is prevalent in both children and adults, and in both genders . The primary cause of gingivitis is plaque accumulation due to poor oral hygiene; however, gingivitis may result from many varied aetiological factors. Gingivitis is characterized by red, swollen, spongy gums that bleed easily . Current conventional treatment of gingivitis involves removal of plaque and the use of an antimicrobial mouthwash. Mouthwashes containing chlorhexidine gluconate are most commonly prescribed, however these have certain adverse effects. Ora-saltsTM is a commercially available mouthwash composed of natural sea salt, Arnica montana 30 centesimal (C), Echinacea angustifolia 30C, Staphisagria 30C, Phosphorus 30C, Hepar sulph 30C, cinnamon and liquorice. To date there is no research on the use of OrasaltsTM in the treatment of gingivitis. The aim of this study is to determine the efficacy of OrasaltsTM in the treatment of gingivitis using the Modified Gingival Index (MGI) and the Quantitative Gingival Bleeding Index (QGBI).

DETAILED DESCRIPTION:
The research will involve a randomised, double blind, controlled, 8 day study, using matched pairs. The study will take place at the Homoeopathy Health Centre at the University of Johannesburg. The research sample will consist of 40 participants aged between 18 to 70 years who have gingivitis; recruited by means of an advertisement placed at the University of Johannesburg and at a private dental practice with relevant permission given. On day 0 of the study potential participants will be requested to sign the Participant Information and Consent Form, and will be screened using a Screening Questionnaire to evaluate if they meet the inclusion criteria. Those participants who qualify will be invited to participate in the study. The researcher will perform the first clinical assessment on each participant on day 0, using the Modified Gingival Index (MGI) and vital signs will be recorded. Participants will be supplied with one container of 120g containing either OrasaltsTM or the control, consisting of natural unmedicated sea salt. The participants will be supplied with the Quantitative Gingival Bleeding Index (QGBI); they will be requested to complete it on days 1 to 7 of the study, grading the response of their gingivitis throughout the study. They will be requested to use the supplied mouthwash twice a day for 7 days. Participants will be supplied with a leaflet informing them how to use the mouthwash and on the practice of good oral hygiene. Participants will be asked to return on day 8 of the study, where they will return with the completed QGBI form grading the response of their gingivitis. And a second assessment using the MGI will be performed by the researcher, and vital signs will be recorded. Data obtained will be statistically analysed by means of essential data assessment which will determine whether parametric or non-parametric tests will be utilised. A possible outcome of this study is to demonstrate that OrasaltsTM may be effective in the treatment of gingivitis, providing an alternative treatment option for this condition. This will open up the field for further research.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 18 and 70; and
* Have active gingivitis at the time of the study including at least 3 of the following symptoms: red, swollen, and spongy gums; gums that bleed spontaneously or after brushing, eating or touching of the gums; having bad breath; sensation of tingling or itching of the gums; and the presence of pus in the pockets between teeth

Exclusion Criteria:

* • Present with any relevant systemic diseases which are known to cause gingivitis such as conditions affecting the immune system, including autoimmune conditions (Sjögrens syndrome, rheumatoid arthritis, systemic lupus erythematosus, diabetes mellitus etc.) and immune deficiencies such as HIV and AIDS, mental health diseases (such as anxiety or depression), malignancy, thyroid conditions, xerostomia, nutritional deficiencies and uncontrolled hypertension

  * Are taking antibiotics or anti-inflammatory drugs during or for 1 month prior to the study onset
  * Have a known allergy to cinnamon or liquorice; and/or
  * Are taking Warfarin or other blood thinning medication Participants will be requested not to make use of any other medication/mouthwashes to treat their gingivitis for the duration of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Modified Gingival Index (MGI) | 8 days
  MGI is a non-invasive method, used by the researcher, to assess inflammation of the gingiva in all 40 participants, at each consultation.

SECONDARY OUTCOMES:
Quantitative Gingival Bleeding Index (QGBI) | 8 days
  QGBI will be used by the participants to rate gingival bleeding on a daily basis.

CONTACTS AND LOCATIONS:
Overall Officials: Radmila Razlog, MTechHom, Study Director — University of Johannesburg
Locations (1):
- University of Johannesburg, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No